CLINICAL TRIAL: NCT01261182
Title: Study of School Feeding Programs' Impact on Anemia Status in Pre-adolescent Girls and Other Vulnerable Household Members in a Cluster-Randomized Trial in Uganda
Brief Title: Targeting School Feeding Programs at Vulnerable Sub-Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Makerere University (Other); World Bank (Other); United Nations World Food Programme (WFP) (Other); UNICEF (Other)
Responsible Party: Marie Ruel/Director, IFPRI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WB-7135830
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Malnutrition; Cognition
Keywords: Malnutrition; School feeding; Infant nutrition; Mother's nutrition; Fortified food; Anemia; Cluster randomized controlled trials; Effectiveness; Impact evaluation studies; Uganda
MeSH Terms: conditions — Malnutrition; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- In School Feeding (Experimental)
  Interventions: Other: In School Feeding
- Take Home Rations (Experimental)
  Interventions: Other: Take Home Rations
- Control (No Intervention)

INTERVENTIONS:
Other: In School Feeding — The intervention provides meals consisting of 1049 kcals of energy, 32.6 gm protein, and 24.9 gm fat per child per school day and meet at least two thirds of the child's daily vitamin and mineral requirements, including 99 percent of iron requirements. SFP delivers these nutrients in the form of a fortified corn-soy porridge around mid-morning and beans and maize meal or rice at lunch.
  Arms: In School Feeding
Other: Take Home Rations — The rations provided in the intervention are equal in size and composition to the food received in the in-school feeding intervention, but are provided to households once per month.
  Arms: Take Home Rations

SUMMARY:
School feeding programs provide students meals conditional on school attendance, which can have impacts on school participation, cognition and learning, and nutritional outcomes. Although the literature on impacts of school feeding programs is substantial, high quality studies with evaluation designs that provide causal impact estimates are relatively few. Thus program impacts on educational, cognitive and nutritional outcomes are not well-understood, particularly in a field setting. Nutritional impacts in particular are questionable, which may be a result program design. Most studies provide only small transfers to children and examine average macro-nutrient effects of the transfer on the treated children, thus it is not surprising that detection of nutritional gains has been minimal.

This study is a cluster-randomized evaluation of a school feeding program administered by the World Food Programme in the Northern Ugandan Districts of Lira and Pader. The program provides substantially larger food rations than most programs (representing 1/3 of children's daily caloric needs and 99% of iron intake requirements).

The key research objectives are:

1. Impact on the treated: Assess the effectiveness of the program at improving nutritional status, education and cognitive and learning outcomes for school-age children, with particular attention to the anemia status of older school-age girls .
2. Impact on untreated but nutritionally vulnerable sub-groups: Assess the effectiveness of the program at reducing anemia prevalence in mothers and younger siblings.
3. Optimal program design: Assess the differential impacts of a program in which children are fed at school compared with one in which they are given dry rations to bring home.

ELIGIBILITY:
Inclusion Criteria:

* School age children

Exclusion Criteria:

-

Ages: 6 Years to 13 Years | Sex: All
Age Groups: Child
Enrollment: 2083 (Actual)

PRIMARY OUTCOMES:
Mothers' and Children's Nutritional Status | 15 months

SECONDARY OUTCOMES:
Cognitive Performance | 15 months
School achievement | 15 months
School Participation | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Ruel, PhD, Principal Investigator — IFPRI
Locations (2):
- Uganda (2):
  - Lira District, Lira
  - Pader District, Pader

REFERENCES:
- [Derived] Adelman S, Gilligan DO, Konde-Lule J, Alderman H. School Feeding Reduces Anemia Prevalence in Adolescent Girls and Other Vulnerable Household Members in a Cluster Randomized Controlled Trial in Uganda. J Nutr. 2019 Apr 1;149(4):659-666. doi: 10.1093/jn/nxy305. PMID 30926996